CLINICAL TRIAL: NCT00246831
Title: Brain Networks Responsible for Self-Agency: An fMRI Study
Brief Title: Brain Networks Responsible for Self-Agency
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060023; 06-N-0023
Record Dates: First submitted 2005-10-29; First posted 2005-10-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-10-28

CONDITIONS: Brain
Keywords: fMRI; Self-Agency; Functional Magnetic Resonance Imaging (fMRI); Voluntary Movement; Healthy Volunteer; HV

SUMMARY:
This study will examine how people consider their actions to be under their own control or not. The term to describe this feeling of being in control of one's own actions is called "agency." The sense of agency becomes impaired in disorders such as schizophrenia, in which people may feel, for example, as if someone else is controlling their thoughts.

Healthy, right-handed normal volunteers 18 years of age and older may be eligible for this study. Candidates are screened with a medical history, neurological examination, pregnancy test for women of childbearing age, and magnetic resonance imaging (MRI) scan. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. During the procedure, the subject lies on a table that can slide in and out of the scanner (a metal cylinder surrounded by a magnetic field) and may be asked to lie still for up to 30 minutes at a time.

Participants undergo functional MRI (fMRI). This procedure is the same as a regular MRI, except it is done while the subject performs tasks. This enables researchers to learn about changes in brain regions involved in those tasks. The fMRI scan for this study takes about 90 minutes.

Before beginning the fMRI procedure, subjects receive training using a Cyber glove device. This device allows the researchers to measure the subject's finger movements and display them on a screen for the subject to view. The subjects are asked to make hand movements by slowly opening and closing the hand while watching the computer displaying an artificial hand. During the movements, the subjects' level of control is adjusted and they are asked to describe how much control they think they have over the hand on the screen. When the subjects become comfortable using the Cyber glove, they enter the MRI scanner to begin the test scan.

For the fMRI, subjects are given visual instruction on when to begin opening and closing their right hand. They move continuously for a 30-second block and then have a 20-second rest period. This is repeated, with subjects provided different levels of control over the displayed hand in each block. The entire test consists of four runs, each run consisting of 12 blocks lasting about 10 minutes. When the fMRI scanning is finished, the brain is scanned once more using regular MRI.

DETAILED DESCRIPTION:
OBJECTIVE:

The purpose of this study is to identify structural brain regions, using a block design blood oxygenation level-dependent functional magnetic resonance imaging (BOLD-fMRI), which are differentially activated based on the sense of self-agency felt by making simple finger movements. We will compare the activations of healthy volunteers with patients diagnosed with a functional movement disorder (FMD) who we hypothesize will have an impaired sense of volition.

STUDY POPULATION:

We intend to use 25 right-hand dominant, adult healthy volunteers for comparison with 50 patients diagnosed with a FMD. We also wish to study an additinal 5 patients witha complete or near-complete sensory neuropathy.

DESIGN:

The sense of self-agency (SA) will be modulated using a visual task-based stimulus asking subjects to manipulate the position of an artificial hand projected onto a display in the magnetic resonance imaging (MRI) scanner. Subjects will use their own right hand to make slow sequential finger movements which will be represented visually with the aid of a Cyberglove. During a behavioral training phase, subjects will practice using the apparatus. The level of control will be randomly changed to one of five states: 100% control, 75%, 50%, 25%, or random/no control. After subjects are comfortable with the apparatus and endorse SA over the displayed hand, they will undergo fMRI scanning. FMD patients who do not wish to participate in the fMRI portion of the study may still participate in the behavioral testing portion.

The imaging phase of the experiment will have five sets of 6 minute scanning sessions where the subject is instructed to slowly open and close sequential fingers of their right hand. The level of control will be changed pseudo-randomly throughout the scan sessions. A control contrast consisting of the subject observing a moving hand will also be integrated into the blocks. An additional control contrast involving the subject moving their hand without visual feedback will also be included. These contrasts will serve in the analysis phase to help eliminate hemodynamic activity related to visual-motor feedback. At the completion of fMRI scanning, a baseline high-resolution MRI T1 scan will be obtained for anatomic localization and co-registration. At the completion of the imaging portion, subjects will also be asked to report the percentage of control they subjectively feel over the displayed hand using a final data set for behavioral testing.

OUTCOME MEASURES:

The primary outcome of this study is the difference in activation of brain structures in response to a loss of SA between FMD patients, sensory neuropathy patients, and healthy controls. In particular, we are interested in the presence of any differential activation in the dorsolateral prefrontal cortex, insula, inferior parietal lobes, pre-supplementary motor association cortex (pre-SMA), and/or the anterior cingulate which may occur as SA is increased or decreased. A secondary analysis will utilize the individual subject perceptions of percent control during the behavioral training phase as the regressors for activation rather than the objective control settings.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects age 18 and older.
* Subjects must be right-hand dominant (For healthy controls).
* Patients diagnosed with a probable or definite functional movement disorder by an HMCS physician or diagnosed with complete or near-complete sensory neuropathy.
* Subjects willing to abstain from caffeine or alcohol for 48 hours prior to the fMRI scanning.

EXCLUSION CRITERIA:

* Subjects with any abnormal findings on neurological exam.
* Subjects with a positive urine pregnancy test.
* Subjects who are pregnant.
* Subjects with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan.
* Subjects with metallic dental fillings which are likely to cause MRI artifacts.
* Subjects with any history of brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies.
* Subjects with any history of a severe medical condition, such as cardiovascular disease, which would prevent them from lying flat for up to 120 minutes.
* Subjects without the capacity to give informed consent.
* Subjects with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 60 minutes.
* Patients with excessive movements at rest.
* Patients with symptom remission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-10-27; Study Completion 2008-10-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gallagher S. Philosophical conceptions of the self: implications for cognitive science. Trends Cogn Sci. 2000 Jan;4(1):14-21. doi: 10.1016/s1364-6613(99)01417-5. PMID 10637618
- [Background] Kircher TT, Leube DT. Self-consciousness, self-agency, and schizophrenia. Conscious Cogn. 2003 Dec;12(4):656-69. doi: 10.1016/s1053-8100(03)00071-0. PMID 14656508
- [Background] Blakemore SJ, Frith CD, Wolpert DM. The cerebellum is involved in predicting the sensory consequences of action. Neuroreport. 2001 Jul 3;12(9):1879-84. doi: 10.1097/00001756-200107030-00023. PMID 11435916